CLINICAL TRIAL: NCT07217366
Title: Testing a Speech-to-text Tool for Heart Failure Patient-Reported Data
Brief Title: Speech-to-text Tool for Heart Failure Patient-Reported Data
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Alexander Sandhu, Assistant Professor of Medicine, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 79867
Record Dates: First submitted 2025-10-13; First posted 2025-10-16 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Heart Failure
Keywords: Artificial intelligence; Speech-to-text; Patient-reported data; Digital health; Patient self-care
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AI Voice Assistant (Experimental): Participants in the AI Voice Assistant arm will complete two activities: (1) an interaction with the AI Voice Assistant tool and (2) Paper survey that includes the same questions asked by AI voice assistant. Half of the participants will use the AI Voice Assistant first, while the other half will begin with the paper survey.
  Interventions: Other: Artificial intelligence speech-to-text tool

INTERVENTIONS:
Other: Artificial intelligence speech-to-text tool — Pilot testing of speech-to-text tool using artificial intelligence

SUMMARY:
The goal of this study is to see whether this type of Artificial Intelligence (AI) Voice Assistant can reliably capture patient-reported health information to support communication between patients and their healthcare team.

ELIGIBILITY:
Inclusion Criteria:

* Adults with heart failure receiving cardiology care at Stanford University

Exclusion Criteria:

* Diminished decision-making capacity
* Inability to understand and communicate in English sufficiently to complete study procedures
* Inability to complete study procedures to the best of the participant's and investigator's knowledge
* Any disorder or condition that, in the opinion of the investigator would pose a risk to participant safety or interfere with the study evaluation, procedures or completion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Accuracy of AI Voice Assistant Compared With Expert Extraction | ~3 months
  Agreement between AI-generated summaries and expert-reviewed responses (study staff extraction of participants' responses from audio recordings). The responses will be scored on a numerical scale, ranging from 0-17 points with higher points representing greater accuracy of the AI-generated summaries compared to expert-reviewed responses.

SECONDARY OUTCOMES:
Usability of AI Voice Assistant | ~3 months
  Measured using the System Usability Scale (SUS), a validated 10-item questionnaire rated on a 5-point Likert scale, with total scores ranging from 0-100
Agreement between AI Voice Assistant Compared With Patient Self-Reported Written Responses | ~3 months
  We will compare agreement the AI Voice Assistant summary to patient-reported responses on the same data elements, including vital signs (heart rate, blood pressure, weight) and 14 symptom and health status questions. The responses will be scored on a numerical scale, ranging from 0-17 points with higher points representing higher agreement of the AI-generated summaries compared to expert-reviewed responses.
Symptom Scores | ~3 months
  Symptom scores based on the responses to questions obtained from AI Voice Assistant and written responses
Qualitative Feedback | ~3 months
  Open-ended questions inquiring about participants' likes, dislikes, and suggestions for improvements

OTHER OUTCOMES:
Time | ~3 months
  Time to complete AI Voice Assistant call and Paper Survey

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Sandhu, MD, MS, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Investigators can provide documents including the study protocol, study analysis plan, and informed consent form of the study to researchers who request the information
Supporting Information: Study Protocol
Time Frame: December 2025-December 2026